CLINICAL TRIAL: NCT05170815
Title: Clariance Registry of ERISMA® and Idys® Devices
Brief Title: Clariance ErYs Registry
Acronym: ErYs
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Clariance (Industry)
Responsible Party: Sponsor
Other Study IDs: CSS-2021-01
Record Dates: First submitted 2021-11-25; First posted 2021-12-28 (Actual); Last update posted 2022-07-22 (Actual); Status verified 2022-07

CONDITIONS: Spine Degeneration; Spine Spondylosis Thoracic; Spinal Deformity; Spinal Tumor; Spinal Fracture
MeSH Terms: conditions — Spinal Cord Neoplasms; Spinal Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (11):
- ERISMA® LP/LP EVO: 120 subjects with ERISMA® LP/LP EVO implant
  Interventions: Procedure: Spine surgery
- ERISMA® Deformity: 120 subjects with ERISMA® Deformity implant
  Interventions: Procedure: Spine surgery
- ERISMA® MIS: 120 subjects with ERISMA® MIS implant
  Interventions: Procedure: Spine surgery
- Idys® TLIF PEEK: 50 subjects with Idys® TLIF PEEK implant
  Interventions: Procedure: Spine surgery
- Idys® TLIF TiVAC: 50 subjects with Idys® TLIF TiVAC implant
  Interventions: Procedure: Spine surgery
- Idys® TLIF 3DTi: 50 subjects with Idys® TLIF 3DTi implant
  Interventions: Procedure: Spine surgery
- Idys® ALIF PEEK: 50 subjects with Idys® ALIF PEEK implant
  Interventions: Procedure: Spine surgery
- Idys® ALIF TiVAC: 50 subjects with Idys® ALIF TiVAC implant
  Interventions: Procedure: Spine surgery
- Idys® ALIF 3DTi: 50 subjects with Idys® ALIF 3DTi implant
  Interventions: Procedure: Spine surgery
- Idys® ALIF ZP 3DTi: 50 subjects with Idys® ALIF ZP 3DTi implant
  Interventions: Procedure: Spine surgery
- Idys® LLIF 3DTi: 50 subjects with Idys® LLIF 3DTi implant
  Interventions: Procedure: Spine surgery

INTERVENTIONS:
Procedure: Spine surgery — Implantation of spine Interbody Fusion Devices and/or Posterior fixation System.

SUMMARY:
International, prospective, single arm, multicenter and observational Post-Market Clinical Follow-up (PMCF).

The overall objective of this study is to collect preoperative, intraoperative and postoperative (at 9 weeks, 6 months, 1 year and 2 years) data on the clinical complications and functional outcomes of the study devices to demonstrate safety and performance in a real-world setting.

The primary objective is to demonstrate that the use of the study devices is safe.

The secondary objective is to demonstrate that the use of the study devices decreases the pain, and improves the quality of life and the daily activities of the subjects.

ELIGIBILITY:
Inclusion Criteria:

* Considered as adult in the respective geography (18 years old or older for France and 21 years old or older for United-States).
* Indicated for treatment with one or more commercially available sponsor spine device included into the study.
* For France only, affiliated with or beneficiary of a social security scheme.

Exclusion Criteria:

* Subjects who are not able to comply with the study procedures based on the judgment of the investigator (e.g., inability to comprehend study related questions, inability to keep scheduled assessment times).
* Subjects who are considered as vulnerable: minor, pregnant woman or people under legal protection (guardianship or curatorship).
* Contraindicated for spine surgery utilizing a commercially available sponsor spine device.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with thoracolumbar disease, and who require spine surgery with Interbody Fusion Device and/or Posterior fixation System
Sampling Method: Probability Sample
Enrollment: 760 (Estimated)
Dates: Start 2022-01-17 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Revision rate | Year 2
  Revision (each time a primary study implant is removed during an additional necessary surgery) rates, as a percentage of the total of cases per primary study device.

SECONDARY OUTCOMES:
Back & Leg Pain Visual Analog Score (VAS) | Pre-op; Week 9; Month 6; Year 1; Year 2
  Self-report scale consisting in a 10-centimeter horizontal line with each end being an extreme label of the pain or discomfort experienced by the subject. The extreme labels are "no pain" (corresponding to the scale of 0) and "the worst pain imaginable" (corresponding to the scale of 100).
Oswestry Disability Index (ODI) | Pre-op; Week 9; Month 6; Year 1; Year 2
  Self-report scale with 10 items each which 6 statements referring to the subject's life in different scenarios. The answers are scored on a 0 - 5 points scale that is then transformed to result in a score that ranges from 0% (indicating least disability) to 100% (indicating most disability).
Self-report multipurpose short-form (SF-12v2®) | Pre-op; Week 9; Month 6; Year 1; Year 2
  The SF-12v2® measures eight components of general health: physical functioning, role limitations due to physical health problems, bodily pain, general health, vitality (energy/fatigue), social functioning, role limitations due to emotional problems and mental health (psychological distress and psychological wellbeing).
Subject's Satisfaction | Week 9; Month 6; Year 1; Year 2
  Five questions regarding the surgery outcomes, if the subject would recommend the surgery to family members and if the subject would still undergo the surgery. Each answer indicates a different level of satisfaction.
Radiological parameter: bony fusion | Week 9; Month 6; Year 1; Year 2
  Evaluation of the interbody fusion from either X-rays or CT-scan images.
Adverse Events | Through study completion, an average of 2 years
  Number of untoward medical occurrences, unintended diseases or injuries, or untoward clinical signs (including abnormal laboratory findings) in subjects , users or other persons, whether or not related to the investigational medical device and whether anticipated or unanticipated. May be serious or not.
Device Deficiencies | Through study completion, an average of 2 years
  Number of inadequacies of a medical device with respect to its identity, quality, durability, reliability, usability, safety or performance.

CONTACTS AND LOCATIONS:
Locations (1):
- Santy Orthopedic Center, Lyon, France